CLINICAL TRIAL: NCT03227055
Title: Cardiovascular Comorbidity in Children With Chronic Kidney Disease: Identification of Novel Biomarkers and Therapeutic Targets
Brief Title: Cardiovascular Comorbidity in Children With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tain, You-Lin, Professor, Chang Gung Memorial Hospital
Other Study IDs: 201601181A3
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Childhood Chronic Kidney Disease
Keywords: Arterial stiffness, children, chronic kidney disease, hypertension, microRNA
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, urine, and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD: Children and adolescents with stage G1-G4 CKD, age 3 to 18 yr

SUMMARY:
This 3-year study will systematically evaluate the prevalence, clinical symptoms, and progression of CV and kidney disease and assess the impact of potential genetic, pharmacological, behavior, and environmental risk factors in a prospective cohort with a sample size of 125 aged 3-18 years children with stage G1-G4 chronic kidney disease (CKD). Measurements of morphological (e.g., LVMI & cIMT) and functional characteristics (e.g., FMD & PWV) of the cardiovascular system and 24hr ABPM profile will serve as surrogate end points for CV comorbidity in this study. Possible associations of these end points with multiple molecular (ADMA & urine exosome miRNA), perceived value and behavior (EQ-5D-Y), pharmacological (NHIRD and CGRD), and environmental risk factors (patient and family survey) will be explored.

DETAILED DESCRIPTION:
Taiwan has the highest incidence and prevalence rates of end-stage renal disease all over the world. Chronic kidney disease (CKD) becomes a global public health burden, which can begin in earliest childhood. CKD in childhood differs from that in adults. Congenital anomalies of the kidney and urinary tract (CAKUT) is the leading cause of childhood CKD. Children with CKD due to CAKUT have the highest risk of having a genomic imbalance. Thus, early identification of genotype-phenotype correlations to develop novel therapeutic approaches might reduce the heavy burden of CKD for the future of Taiwan.

Study design:

1. A 3-year prospective cohort study.
2. Sample size: 125 children and adolescents with stage G1-G4 CKD, age 3 to 18 yr, and 30 controls.

4. Measurement: Measurements of morphological (e.g., LVMI & cIMT) and functional characteristics (e.g., FMD & PWV) of the cardiovascular system and 24hr ABPM profile will serve as surrogate end points for CV comorbidity in this study. Possible associations of these end points with multiple molecular (ADMA & urine exosome miRNA), perceived value and behavior (EQ-5D-Y), pharmacological (NHIRD and CGRD), and environmental risk factors (patient and family survey) will be explored.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents with stage G1-G4 CKD

Exclusion Criteria:

* current pregnancy
* inability to complete major data collection
* kidney transplant
* cancer

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 125 children and adolescents with stage G1-G4 CKD and 30 controls.
Sampling Method: Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2016-12-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Hypertension | 1 year
  Abnormal ABPM profile

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No